CLINICAL TRIAL: NCT01534117
Title: Platelet Function Analysis in Head Trauma: ASA/CLOPIDOGREL
Brief Title: Platelet Function Analysis in Head Trauma: ASA/Plavix
Acronym: ASA/Plavix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang, Steve S., M.D. (Individual)
Collaborators: Santa Barbara Cottage Hospital (Other); Accumetrics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: ASA/Plavix/Platelets_SBCH
Record Dates: First submitted 2012-02-08; First posted 2012-02-16 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Head Injury Trauma Blunt
MeSH Terms: interventions — Platelet Count; Deamino Arginine Vasopressin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Platelets/DDAVP (Active Comparator): Fall on ASA/Plavix that sustained head trauma requiring administration of platelets and/or DDAVP
  Interventions: Biological: Platelets; Drug: DDAVP
- No Platelets (No Intervention): Those that sustain head trauma NOT requiring platelet transfusion. The investigators are evaluating platelet function in those not requiring platelet transfusion

INTERVENTIONS:
Biological: Platelets — 1 unit of platelets
  Arms: Platelets/DDAVP
Drug: DDAVP — Desmopressin 0.3mcg/kg IV x 1
  Arms: Platelets/DDAVP

SUMMARY:
The investigators are assessing the platelet function analysis of those who sustained significant head trauma while on aspirin or plavix and to assess if any qualitative difference is obtained if platelets are administered.

DETAILED DESCRIPTION:
The platelet function analyzer VerifyNow® P2Y12 uses ADP as agonists to induce platelet activation and ascertain the level of platelet function impaired by these medications. VerifyNow® Aspirin Assay utilizes arachidonic acid as the agonist to measure platelet function specifically along this pathway. Our research question for this study is as follows:

Does the administration of desmopressin (DDAVP) and/or the transfusion of platelets in patients with head trauma reverse the platelet inhibition caused by Aspirin and/or Plavix? The investigators hypothesize that with the administration of platelets and/or DDAVP that there is a reversal of the inhibition.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18yrs
2. Must be a trauma patient with blunt head trauma.
3. Must be on Aspirin and/or Plavix
4. Subject or Legally Authorized Representative (LAR) (per Heath and Safety Code, Sections 24170 to 24179.5) must sign study consent within 4 hours from the first blood draw. (If this criterion is not met the initial blood draw must be destroyed and NOT run for study results).

Exclusion Criteria:

1. Hemoglobin ≤ 10 GM/DL
2. Platelet Count ≤ 150 K/MCL
3. Pregnant Females
4. Subjects on Warfarin, Heparin or Enoxaparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-10; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Platelet inhibition | 8 hours
  We are measuring platelet inhibition using the verify now platelet function analyzer

CONTACTS AND LOCATIONS:
Overall Officials: Steve S Chang, MD, Principal Investigator — Santa Barbara Cottage Hospital
Locations (1):
- Santa Barbara Cottage Hospital, Santa Barbara, California, United States